CLINICAL TRIAL: NCT05322434
Title: The Effect Of Online Breastfeeding Counseling Given At The Post-Birth Period On Breastfeeding Behavior
Acronym: Breastfeed
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Beyza Akturk, Midwife, Marmara University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Breastfeeding counseling
Record Dates: First submitted 2022-03-14; First posted 2022-04-11 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Breastfeeding; Breastfeeding Support
Keywords: Postpartum period; Breastfeeding; time to start solid food; online; consultancy
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): Postpartum breastfeeding training, which is routinely done immediately after birth, and breastfeeding counseling will be provided in the 1st, 2nd, 4th and 6th months after birth.
  Interventions: Other: The Effect Of Online Breastfeeding Counseling Given At The Post-Birth Period On Breastfeeding Behavior
- control group (No Intervention): Postpartum breastfeeding education will be given routinely immediately after birth.

INTERVENTIONS:
Other: The Effect Of Online Breastfeeding Counseling Given At The Post-Birth Period On Breastfeeding Behavior — The aim of the study is to investigate breastfeeding behavior and initiation of solid food by giving breastfeeding counseling to women within the framework of the Health Belief Model for 6 months from birth.
  Arms: experimental group

SUMMARY:
The World Health Organization and the United Nations Children's Fund recommend that every baby be fed with breast milk alone from birth to 6 months, then with additional foods; recommends continuation of breastfeeding until at least 2 years of age. It has been reported that with the spread of breastfeeding, 823,000 child and 20,000 maternal deaths can be prevented and 300 billion dollars of economic savings can be made every year in the world. The COVID 19 pandemic, which has been affecting the whole world for the last two years, has led to changes in the field of consultancy as well as in all areas. Counseling has created a tendency to be given online due to the rapid spread of the virus, the fact that it is deadly, and the increased risk in closed areas.

There has been a great deal of interest in the subject of breastfeeding behavior in the literature, but it has been observed that there is not enough research on breastfeeding counseling given online. In this study, breastfeeding behavior of mothers in the first six months and the duration of starting solid food will be investigated.

DETAILED DESCRIPTION:
Breastfeeding has a biological and emotional effect on mother and baby, and has many immunological, psychological, social and economic benefits for both mother and baby. The content of breast milk is regulated according to the needs of the baby, regardless of the mother's diet. The importance of breastfeeding in laying the foundations of a healthy life is indisputable.The World Health Organization and the United Nations Children's Fund recommend that every baby be fed with breast milk alone from birth to 6 months, then with additional foods; recommends continuation of breastfeeding until at least 2 years of age. It has been reported that with the spread of breastfeeding, 823,000 child and 20,000 maternal deaths can be prevented and 300 billion dollars of economic savings can be made every year in the world.

WHO for the protection, promotion and dissemination of breastfeeding; It recommends the full adoption of the 'International Law on the Marketing of Breastmilk Substitutes (Food Code)' adopted in 1981, the widespread implementation of the 'Ten Steps to Successful Breastfeeding' principles within the scope of the Baby-Friendly Health Institutions Program, and increasing community-based support such as mother support groups and trainings. In addition, it is recommended to provide counseling and support about breastfeeding at every opportunity where the baby and parents can be contacted, such as antenatal-postnatal follow-ups, child health follow-ups and applications due to illness. Eker and Yurdakul stated in their study that it is the midwife and nurse's responsibility to provide continuous monitoring and control of mothers in the postpartum period, and they reported that providing breastfeeding education and counseling after discharge positively affects breastfeeding success.The COVID 19 pandemic, which has been affecting the whole world for the last two years, has led to changes in the field of consultancy as well as in all areas. Counseling has created a tendency to be given online due to the rapid spread of the virus, the fact that it is deadly, and the increased risk in closed areas.

In this study, breastfeeding counseling will be given to women in the postpartum period online in our country, where early cessation of breastfeeding and early initiation of complementary foods is a serious problem. There has been a great deal of interest in the subject of breastfeeding behavior in the literature, but it has been observed that there is not enough research on breastfeeding counseling given online. In this study, breastfeeding behavior of mothers in the first six months and the duration of starting solid food will be investigated.Data will be obtained using the Data Collection Form and the Breastfeeding Self-Efficacy Scale Short Form. Data Collection Form; It was created as a result of scanning and examining the relevant literature by the researcher, which includes socio-demographic characteristics. This form will be applied after completing the informed consent form and obtaining the participant's consent. Breastfeeding Self-Efficacy Scale Short Form; The Breastfeeding Self-Efficacy Scale was first developed by Dennis and Faux as a 33-item scale. This scale evaluates the mothers' feeling of self-sufficiency regarding breastfeeding.

The data obtained from the research will be statistically analyzed using the International Business Machines Statistical Package for Social Sciences Subscription trial version in computer environment. The descriptive characteristics of the participants will be evaluated by number, percentage, lowest and highest values, mean, standard deviation. Breastfeeding Self-Efficacy Scale and ANOVA, t-Test, Mann Whitney U Test, Kruskal Wallis Test, Mean, Standard Deviation will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* volunteer,
* be between 18-45 years old,
* Not having a condition that prevents breastfeeding,
* Being primiparous,
* be a smart phone

Exclusion Criteria:

* The form is not completely filled

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Postpartum women
Enrollment: 94 (Estimated)
Dates: Start 2023-05-01 (Estimated); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
The Effect Of Online Breastfeeding Counseling Given At The Post-Birth Period On Breastfeeding Behavior | 7 months
  The minimum score that can be obtained from the breastfeeding self-efficacy scale is 14, and the maximum is 70. A high score is an indicator of high breastfeeding self-efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Meltem Demirgöz Bal, Assoc. Dr., Study Director — Head of Department of Midwifery at Marmara University

IPD SHARING:
Plan to Share IPD: No